CLINICAL TRIAL: NCT04294160
Title: A Phase Ib, Multicenter, Open-label Dose Escalation and Expansion Platform Study of Select Drug Combinations in Adult Patients With Advanced or Metastatic BRAF V600 Colorectal Cancer
Brief Title: A Study of Select Drug Combinations in Adult Patients With Advanced/Metastatic BRAF V600 Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision of early termination was made due to business reasons, and was not based on any safety concerns for any of the treatment combinations.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CADPT01C12101
Record Dates: First submitted 2020-03-02; First posted 2020-03-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: BRAF V600 Colorectal Cancer
Keywords: Phase Ib, BRAF-mutated, BRAF V600E, BRAF V600D, BRAF V600K, colorectal cancer, colon cancer, rectal cancer, metastatic, BLRM with EWOC
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasm Metastasis | interventions — dabrafenib; trametinib; naporafenib; spartalizumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dabrafenib + LTT462 backbone arm 1 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer
  Interventions: Drug: Dabrafenib; Drug: LTT462
- Dabrafenib + LTT462 + trametinib triplet arm 1 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer
  Interventions: Drug: Dabrafenib; Drug: LTT462; Drug: Trametinib
- Dabrafenib + LTT462 + LXH254 triplet arm 2 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer - Arm is closed for further enrollment.
  Interventions: Drug: Dabrafenib; Drug: LTT462; Drug: LXH254
- Dabrafenib + LTT462 + TNO155 triplet arm 3 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer
  Interventions: Drug: Dabrafenib; Drug: LTT462; Drug: TNO155
- Dabrafenib + LTT462 + spartalizumab triplet arm 4 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer - Arm is closed for further enrollment.
  Interventions: Drug: Dabrafenib; Drug: LTT462; Biological: Spartalizumab
- Dabrafenib + trametinib + TNO155 triplet arm 5 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: TNO155
- Dabrafenib + LTT462 + Tislelizumab triplet arm 6 (Experimental): dose escalation to determine maximum tolerated dose (MTD)/ Recommended dose (RD) in adult patients with advanced or metastatic BRAF V600 colorectal cancer
  Interventions: Drug: Dabrafenib; Drug: LTT462; Biological: Tislelizumab

INTERVENTIONS:
Drug: Dabrafenib — Capsule for oral use
  Other Names: DRB436, Tafinlar
Drug: LTT462 — Capsule for oral use
  Arms: Dabrafenib + LTT462 + LXH254 triplet arm 2; Dabrafenib + LTT462 + TNO155 triplet arm 3; Dabrafenib + LTT462 + Tislelizumab triplet arm 6; Dabrafenib + LTT462 + spartalizumab triplet arm 4; Dabrafenib + LTT462 + trametinib triplet arm 1; Dabrafenib + LTT462 backbone arm 1
Drug: Trametinib — Tablet for oral use
  Other Names: TMT212, Mekinist
  Arms: Dabrafenib + LTT462 + trametinib triplet arm 1; Dabrafenib + trametinib + TNO155 triplet arm 5
Drug: LXH254 — Tablet for oral use
  Arms: Dabrafenib + LTT462 + LXH254 triplet arm 2
Drug: TNO155 — Capsule for oral use
  Arms: Dabrafenib + LTT462 + TNO155 triplet arm 3; Dabrafenib + trametinib + TNO155 triplet arm 5
Biological: Spartalizumab — Liquid in vial (Concentrate for solution for infusion) for intravenous use
  Other Names: PDR001
  Arms: Dabrafenib + LTT462 + spartalizumab triplet arm 4
Biological: Tislelizumab — Liquid in vial (Concentrate for solution for infusion) for intravenous use
  Other Names: VDT482, BGBA317
  Arms: Dabrafenib + LTT462 + Tislelizumab triplet arm 6

SUMMARY:
A phase Ib, open-label platform study of select drug combinations chosen in order to characterize safety and tolerability of each treatment arm tested and to identify recommended doses and regimens for future studies.

DETAILED DESCRIPTION:
This is a phase Ib, multi-center, open-label study with multiple treatment arms in adult patients with advanced or metastatic BRAF V600 (E, D, or K) in order to characterize safety and tolerability of each treatment arm tested and to identify recommended doses and regimens for future studies. The open platform design of this study is adaptive to allow removal of combination treatment arm(s) based on emerging data and facilitate introduction of new candidate combinations. The study is comprised of a dose escalation part and may be followed by a dose expansion part for any combination treatment arm.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patients must be willing to undergo a new tumor biopsy at baseline and during on study therapy. Exceptions may be considered after documented discussion with Novartis.
* All patients must have a BRAF V600 mutation confirmed by local assessment.
* Patients with unresectable advanced/metastatic BRAF V600 cancer of the colon or rectum with measurable disease as determined by RECIST v1.1
* Patients must have documented disease progression following, or are intolerant to, 1 or 2 lines of chemotherapy for advanced/metastatic disease

Key Exclusion Criteria:

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in-situ cervical cancer, or other tumors that will not affect life expectancy
* Impairment of gastrointestinal function or gastrointestinal disease that may signficantly alter the absorption of study drugs
* History of or current evidence/risk of retinal verin occlusion or serous retinopathy
* History of or current interstitial lung disease or non-infectious pneumonitis
* Patients with a known history of testing positive for HIV
* Clinically significant cardiac disease at screening
* Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Pregnant or lactating women

Other protocol-defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose limiting toxicities (DLTs) in the first cycle | 30 months
  To characterize safety and tolerability of each treatment arm tested and identify recommended doses (RD) and regimens for future studies
Incidence and severity of AEs and SAEs, including changes in laboratory values, vital signs, and ECGs | 34 months
  To characterize safety and tolerability of each treatment arm tested and identify recommended doses and regimens for future studies
Frequency of dose interruptions | 30 months
  To characterize safety and tolerability of each treatment arm tested and identify recommended doses and regimens for future studies
Frequency of dose reductions | 30 months
  To characterize safety and tolerability of each treatment arm tested and identify recommended doses and regimens for future studies
Dose intensity | 30 months
  To characterize safety and tolerability of each treatment arm tested and identify recommended doses and regimens for future studies

SECONDARY OUTCOMES:
AUClast derived from Serum/plasma concentration of individual investigational drugs within combination treatments | 30 months
  To characterize the PK of each investigational drug within each treatment arm
Best overall response (BOR) | 34 months
  To evaluate preliminary anti-tumor activity of each treatment arm per RECIST v1.1.
Progression free survival (PFS) | 34 months
  To evaluate preliminary anti-tumor activity of each treatment arm per RECIST v1.1.
Overall response rate (ORR) | 34 months
  To evaluate preliminary anti-tumor activity of each treatment arm per RECIST v1.1.
Duration of response (DOR) | 34 months
  To evaluate preliminary anti-tumor activity of each treatment arm per RECIST v1.1.
Disease control rate (DCR) | 34 months
  To evaluate preliminary anti-tumor activity of each treatment arm per RECIST v1.1.
Change from baseline of the PD marker DUSP6 in tumor tissue (dose escalation only) | 30 months
  To evaluate PD effect in their respective combinations in tumor
AUCtau derived from Serum/plasma concentration of individual investigational drugs within combination treatments | 30 months
  To characterize the PK of each investigational drug within each treatment arm
Cmax derived from Serum/plasma concentration of individual investigational drugs within combination treatments | 30 months
  To characterize the PK of each investigational drug within each treatment arm
Tmax derived from Serum/plasma concentration of individual investigational drugs within combination treatments | 30 months
  To characterize the PK of each investigational drug within each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (4):
  - University of California LA Santa Monica Location, Los Angeles, California
  - Massachusetts General Hospital Massachusetts General Hospital, Boston, Massachusetts
  - Sarah Cannon Research Institute SC, Nashville, Tennessee
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (3):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Zoetermeer, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CADPT01C12101 Clinical Trial results Form — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18353
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2873